CLINICAL TRIAL: NCT01460108
Title: Utility of the AeriSeal System in Patients With Advanced Upper Lobe Predominant Emphysema and Collateral Ventilation Assessed by the Chartis System
Brief Title: AeriSeal System in Patients With Advanced Upper Lobe Predominant Emphysema and Collateral Ventilation
Acronym: CV+
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LudwLudwig Boltzmann Institute for COPD and Respiratory Epidemiology (Network)
Responsible Party: Principal Investigator, Arschang Valipour, Ass. Prof. Department of Respiratory and Critical Care Medicine, LudwLudwig Boltzmann Institute for COPD and Respiratory Epidemiology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EK_11_027_0311
Record Dates: First submitted 2011-10-25; First posted 2011-10-26 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Pulmonary Emphysema; COPD; Lung Diseases
Keywords: PLVR; AeriSeal; Treatment; Device; Breathing; COPD; emphysema; polymeric lung volume reduction; heterogeneous; homogeneous; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Emphysema; Pulmonary Disease, Chronic Obstructive; Lung Diseases; Respiratory Aspiration; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AeriSeal System Treatment (Experimental): Candidates for the trial include patients with advanced non-bullous upper lobe predominant emphysema who have a DLco between 20 and 60% predicted and target sites in at least 1 upper lobe. Eligible and consented patients will undergo evaluation with the Chartis System, and only patients found to have significant collateral ventilation will be enrolled.
  Interventions: Device: AeriSeal System

INTERVENTIONS:
Device: AeriSeal System — 20 mL
  Other Names: Emphasemateous Lung Sealant

SUMMARY:
The purpose of this study is to characterize the safety and efficacy of the AeriSeal System in patients with advanced upper lobe predominant emphysema and significant collateral ventilation as determined by the Chartis System.

DETAILED DESCRIPTION:
This is an investigator initiated, open-label, uncontrolled study to prospectively characterize the safety and efficacy of the AeriSeal System in patients with advanced upper lobe predominant emphysema found to have significant collateral ventilation using the Chartis System.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent and to participate in the study
* Diagnosis of advanced emphysema (GOLD Stage III or Stage IV disease)
* Radiologic evidence of non-bullous upper lobe predominant heterogeneous emphysema with at least 2 target sites deemed appropriate for treatment evident by CT imaging
* DLco between 20 and 60% predicted
* Positive Collateral Ventilation as determined by the Chartis® System
* Clinically significant dyspnea (defined as a MRC dyspnea score of 2 or greater at Screening)
* Failure of standard medical therapy to provide adequate relief of symptoms (defined as regular use of standard medication for more than 1 month prior to Screening; standard medications include at least an inhaled beta agonist and inhaled anticholinergic unless medically contraindicated or prior medical failure)
* Significant airflow obstruction as demonstrated by Spirometry 15 minutes after administration of bronchodilator with:
* 5% < FEV1 < 50% predicted using the ATS recommended calculation for expected value
* FEV1/FVC ratio <70%
* Physiological evidence of hyperinflation with Lung volumes (plethysmographic) of:
* TLC > 100% predicted using the ATS recommended calculation for expected value
* RV > 135% predicted using the ATS recommended calculation for expected value
* Six-Minute Walk Test distance ≥ 150 m
* Abstinence from inhaled tobacco use for at least 16 weeks prior to the initial Screening visit until the end of the study
* Female patients are either post-menopausal or surgically sterile. Women with child-bearing potential will not be included in this study

Exclusion Criteria:

* Alpha-1 antitrypsin serum level of < 80 mg/dL (i.e. < 11 micro mol/L) at Screening
* Body mass index < 15 kg/m2 or > 35 kg/m
* Clinically significant asthma, chronic bronchitis or bronchiectasis as determined by the Investigator, or a significant COPD exacerbation within the past 4 months
* Use of systemic steroids > 20 mg/day or equivalent immunosuppressive agents, heparins, oral anticoagulants (e.g., warfarin, dicumarol; note: antiplatelet drugs including aspirin and clopidogrel are permitted) or investigational medications within 4 weeks of Screening
* Allergy or sensitivity to medications required to safely perform AeriSeal System treatment under general anesthesia or conscious sedation
* Participation in an investigational study of a drug, biologic, or device not currently approved for marketing within 30 days prior to the Screening visit
* Prior lung volume reduction surgery, prior lobectomy or pneumonectomy, prior lung transplantation, prior airway stent placement, prior pleurodesis, or prior endobronchial lung volume reduction therapy of any type
* Significant co-morbidity that carries prohibitive risks (e.g., HIV/AIDS, cancer) or is associated with less than 2-year expected survival
* Blood gases and oxygen saturation:

  * SpO2 ≤ 90% on > 4 L/min supplemental O2, at rest
  * PaCO2 ≥ 55mmHg
  * DLCO < 20% or > 60% predicted for patients with heterogeneous emphysema
* Chest CT scan: Presence of any of the following radiologic abnormalities:

  * Pulmonary nodule on CT scan greater than 1.0 cm in diameter (Does not apply if present for 2 years or more without increase in size or if proven benign by biopsy/PET)
  * Giant Bullous Disease
  * Radiologic picture consistent with active pulmonary infection, e.g., unexplained parenchymal infiltrate
  * Significant interstitial lung disease (based upon investigator judgment)
  * Significant pleural disease (based upon investigator judgment)
  * Any condition that the Investigator believes would interfere with the intent of the study or would make participation not in the best interest of the patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Change in Forced Expiratory Volume in one second (FEV1) | 12 Weeks
  Change from baseline in FEV1 measurement after 12 weeks following completion of therapy.

SECONDARY OUTCOMES:
Change in Forced Expiratory Volume in one second (FEV1). | 24 Weeks
  Change from baseline in FEV1 at 24 Weeks following completion of therapy
Change in Forced Vital Capacity (FVC) | 12 Weeks and 24 Weeks
  Change from baseline in FVC at 12 and 24 weeks following completion of therapy.
Change in ratio of Residual Volume to Total Lung Capacity (RV/TLC) | 24 Weeks
  Change from baseline in RV/TLC ratio at 24 weeks following completion of therapy.
Change in distance walked in six minutes (6MWT) | 24 Weeks
  Change from baseline in 6MWT distance at 24 weeks following completion of therapy.
Change in Medical Research Council Dyspnea (MRCD) score | 24 Weeks
  Change from baseline in MRCD score at 24 weeks following completion of therapy
Change in health related quality of life assessment (St. George's Respiratory Questionnaire)(SGRQ) | 24 Weeks
  Change from baseline in disease-specific health related quality of life assessment (SGRQ) at 24 weeks following completion of therapy.
Change in Collateral Ventilation | 24 Weeks
  Change from baseline in collateral ventilation at 24 weeks following completion of therapy as measured by the Chartis System.
Unanticipated Serious Adverse Device Effects (USADEs) | 24 Week
  Record of any/all USADEs up to 24 weeks follwoing completion of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Arschang Valipour, MD, FCCP, Principal Investigator — Ludwig-Boltzmann-Institut für COPD und Pneumologische Epidemiologie
Locations (1):
- Otto-Wagner-Spital, Vienna, Austria